CLINICAL TRIAL: NCT05537181
Title: Evaluation of the Combination Treatment With BTL-899 and HPM-6000UF Devices for Abdominal and Pelvic Floor Muscle Strengthening and Overall Improvement in Quality of Life in Elderly Patients
Brief Title: Combination Treatment With BTL-899 and HPM-6000UF Devices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-899_CTUS500
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Pelvic Floor Disorders
Keywords: core strength; abdominal muscles; pelvic floor muscles; quality of life
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BTL-899; HPM-6000UF Treatments (Experimental): The two devices will be used separately in two different treatments. However one treatment visit can comprise both treatments. The BTL-899 will be applied over the abdomen, and the device will induce visible muscle contractions along with mild heating of the muscles. Four (4) treatments once a week will be delivered. The HPM-6000UF device will induce pelvic floor muscle contractions. Six (6) treatments 2-4 days apart will be delivered.
  Interventions: Device: BTL-899; HPM-6000UF Treatments

INTERVENTIONS:
Device: BTL-899; HPM-6000UF Treatments — The two devices will be used separately in two different treatments. However one treatment visit can comprise both treatments. The BTL-899 will be applied over the abdomen, and the device will induce visible muscle contractions along with mild heating of the muscles. Four (4) treatments once a week will be delivered. The HPM-6000UF device will induce pelvic floor muscle contractions. Six (6) treatments 2-4 days apart will be delivered.

SUMMARY:
This study will evaluate the clinical efficacy of the BTL-899 and HPM-6000UF devices in combination for non-invasive strengthening of the core muscles and overall improvement in quality of life in elderly patients.

DETAILED DESCRIPTION:
The study is a prospective, multicenter single-arm, open-label, interventional study. The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete seven (7) treatment visits and two (2) follow-up visits - 1 month and 3 months after the final treatment.

At the baseline visit, medical history will be assessed. Inclusion and exclusion criteria will be verified, and informed consent will be signed. Digital photographs will be taken, waist circumference will be measured, abdominal muscle strength will be measured with a pressure biofeedback device.

The two devices will be used separately in two different treatments. However one treatment visit can comprise both treatments. The BTL-899 will be applied over the abdomen, and the device will induce visible muscle contractions along with mild heating of the muscles. Four (4) treatments once a week will be delivered. The HPM-6000UF device will induce pelvic floor muscle contractions. Six (6) treatments 2-4 days apart will be delivered. There will be three (3) visits where both treatments will be applied consecutively, starting with BTL-899, followed by the therapy with HPM-6000UF.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged 60 years or older (postmenopause when female),
* BMI ≤35kg/m2 seeking treatment for strengthening their pelvic floor or abdominal muscles
* Subjects should be able to understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form.
* Subjects willing and able to abstain from partaking in any concurrent treatments on abdomen and pelvic floor other than the study procedures during study participation.
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs taken.

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators, and neurostimulators)
* Metal implants in the treated area
* Drug pumps
* Malignant tumor
* Pulmonary insufficiency
* Injured or otherwise impaired muscles in the treated area
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations in the treated area
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Poor healing and unhealed wounds in the treatment area
* Following recent surgical procedures when muscle contraction may disrupt the healing process
* Graves' disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of core muscles strength measured by pressure biofeedback device | 5 months
  Change in core muscles strength measured by pressure biofeedback device
Assessment of subject's quality of life based on Subject Satisfaction and Experience Questionnaire | 5 months
  Change in subject's quality of life based on Subject Satisfaction and Experience

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Plastic Surgical Associates, Fort Collins, Colorado
  - Dermatologic Surgery Specialists, Macon, Georgia
  - Men's Health Boston, Chestnut Hill, Massachusetts